CLINICAL TRIAL: NCT05908708
Title: Title: Closed-loop Medtronic 780G System in Youth With Type 1 Diabetes: AWeSoMe Study Group Prospective Trial
Brief Title: Closed-loop Medtronic 780G System in Youth With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government); Assaf-Harofeh Medical Center (Other Government); Maccabi Healthcare Services, Israel (Other); Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Noah Gruber, Pediatric endocrinologist, Sheba Medical Center
Other Study IDs: SHEBA-22-9609-NG-CTIL
Record Dates: First submitted 2023-05-27; First posted 2023-06-18 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Type 1 Diabetes; Child, Only
Keywords: Technology; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Medtronic 780G® hybrid closed loop — Medtronic 780G® hybrid closed loop system uses the commercial "auto-mode" with an insulin pump and continuous glucose monitoring.

SUMMARY:
The goal of this observational study is to describe data on Israeli children and youth using the 780G system including data regarding glycemic control parameters, various questionnaires, sleep data, bioimpedance measures, and dietary parameters. The main questions it aims to answer are: • whether the 780G system will improve glycemic control • whether the psychosocial aspects will improve. Participants will be followed once connected to 780G, at baseline, one, three, and six months after the connection.

DETAILED DESCRIPTION:
Patients and Methods:

The study population will include individuals with type 1 diabetes ages 7-18 years who are managed by the pediatric diabetes teams from the AWeSoMe Study Group (five pediatric diabetes multidisciplinary clinics in Israel; Dana-Dwek Children's Hospital, Edmond and Lily Safra Children's Hospital, Maccabi National Juvenile Diabetes Center, Shamir Medical Center and Wolfson Medical Center) and who chose to purchase 780G out-of-pocket as part of their diabetes care, or are eligible according to the updated Israeli basket to receive it. The decision to use 780G will be made prior to and independent of their entrance to the study, and will be based on preferences of the patients and their parents.

Study design:

A prospective multi-center study (AWeSoMe Study Group) of type 1 diabetes patients using the closed-loop Medtronic 780G system as compared to their previous treatment regimen.

Data will be collected at 4 timepoints: baseline (at initiation of 780G system), after 1 month, three months and 6 months of the closed-loop Medtronic 780G system usage.

Data collection:

All the data collected are available for healthcare providers (doctors, nurses and dieticians) as part of the routine diabetes clinic visit. The information retrieved from the medical files will include sociodemographic characteristics (current age, sex, socioeconomic position by home address, parent's education level, marital status of parents), anthropometric parameters (height, weight and body mass index), pubertal status, physical activity levels and diabetes-related characteristics. Diabetes-related characteristics: age at diagnosis, autoimmune co-morbidities (thyroid disease and Celiac), glycated hemoglobin (HbA1c) and acute complications (severe hypoglycemic episodes and DKA). Insulin pump and CGM downloaded data retrieved during the 2 weeks prior to the clinic visit: mode of insulin therapy (previous and current), total daily insulin dose (Units/kg/day), total daily carbohydrates (grams/day) and CGM metrics. CGM metrics will include: percent time CGM active, mean glucose level, standard deviation (SD), coefficient of variability (CV), time in range (TIR), time above range (TAR), time below range (TBR) and glucose management indicator (GMI). Closed-loop Medtronic 780G system user evaluation: reason for switching from conventional treatment to closed-loop, automode system exits and patient's/parent's perception of closed-loop system.

In addition to the data mentioned above the following data will be collected:

1. Questionnaires for the:

   1. Patients - the quality of life, anxiety, fear of hypoglycemia - child, diabetes management, and nutrition knowledge in diabetes. All of the questionnaires are validated and were translated into Hebrew using the globally-accepted linguistic validation procedure.
   2. Parents - the quality of life, fear of hypoglycemia - parent, diabetes management, sleep quality, and nutrition knowledge in diabetes. All of the questionnaires are validated and were translated into Hebrew using the globally-accepted linguistic validation procedure.
2. Bioimpedance parameters
3. Diet - nutrition evaluation through 3-daily diet notes
4. Sleep - sleep evaluation through parents' 3-daily sleep diaries

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of type 1 diabetes Diabetes duration ≥ 6 months Routine attendance at clinic visits Initiation of 780G system usage

Exclusion Criteria:

Children under the age of 1 year Children without 780G system

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include individuals with type 1 diabetes ages 1-21 years who are managed by the pediatric diabetes teams from the AWeSoMe Study Group (five pediatric diabetes multidisciplinary clinics in Israel; Dana-Dwek Children's Hospital, Edmond and Lily Safra Children's Hospital, Maccabi National Juvenile Diabetes Center, Shamir Medical Center and Wolfson Medical Center) and who chose to purchase 780G out-of-pocket as part of their diabetes care, or are eligible according to the updated Israeli basket to receive it. The decision to use 780G will be made prior to and independent of their entrance to the study, and will be based on preferences of the patients and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Time spent in range (70-180 mg/dL) as assessed from closed-loop Medtronic 780G system | 0,3 months
  Change in time spent in range (70-180 mg/dL) from baseline to three months of closed-loop Medtronic 780G system
Time spent in range (70-180 mg/dL) as assessed from closed-loop Medtronic 780G system | 0,6 months
  Change in time spent in range (70-180 mg/dL) from baseline to six months of closed-loop Medtronic 780G system

SECONDARY OUTCOMES:
HbA1c as assessed from point-of-care clinic visit | 0, 3 months
  Change in HbA1c from baseline to three months of closed-loop Medtronic 780G system
HbA1c as assessed from point-of-care clinic visit | 0, 6 months
  Change in HbA1c from baseline to six months of closed-loop Medtronic 780G system
Time spent below range (≤ 70 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 3 months
  Change in time spent below range (≤ 70 mg/dL) baseline to three months of closed-loop Medtronic 780G system
Time spent below range (≤ 70 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 6 months
  Change in time spent below range (≤ 70 mg/dL and ≤ 54 mg/dL) baseline to six months of closed-loop Medtronic 780G system
Time spent below range (≤ 54 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 3 months
  Change in time spent below range (≤ 54 mg/dL) baseline to three months of closed-loop Medtronic 780G system
Time spent below range (≤ 54 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 6 months
  Change in time spent below range (≤ 54 mg/dL) baseline to six months of closed-loop Medtronic 780G system
Time spent above range (> 180 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 3 months
  Change in time spent above range (> 180 mg/dL) baseline to three months of closed-loop Medtronic 780G system
Time spent above range (> 180 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 6 months
  Change in time spent above range (> 180 mg/dL) baseline to six months of closed-loop Medtronic 780G system
Time spent above range (> 250 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 3 months
  Change in time spent above range (> 250 mg/dL) baseline to three months of closed-loop Medtronic 780G system
Time spent above range (> 250 mg/dL) as assessed from closed-loop Medtronic 780G system | 0, 6 months
  Delta time spent above range (> 250 mg/dL) baseline to six months of closed-loop Medtronic 780G system
Quality of life - child as assessed by a questionnaire | 0, 6 months
  Change in quality of life - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 5, max score 100; the higher the score, the better quality of life.
Quality of life - parent as assessed by a questionnaire | 0, 6 months
  Change in quality of life - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 37, max score 185; the higher the score, the better quality of life.
Trait anxiety - child as assessed by a questionnaire | 0, 6 months
  Change in trait anxiety - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 20, max score 80; the higher the score, the higher the anxiety.
Fear of hypoglycemia - child as assessed by a questionnaire | 0, 6 months
  Change in fear of hypoglycemia - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 25, max score 100; the higher the score, the higher the fear of hypoglycemia.
Fear of hypoglycemia - parent as assessed by a questionnaire | 0, 6 months
  Change in fear of hypoglycemia - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 25, max score 100; the higher the score, the higher the fear of hypoglycemia.
Diabetes management - child as assessed by a questionnaire | 0, 6 months
  Change in diabetes management - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 20, max score 100; the higher the score, the better the management of diabetes.
Diabetes management - parent as assessed by a questionnaire | 0, 6 months
  Change in diabetes management - baseline to 6 months. A validated questionnaire, as cited in the Reference section. Min score 20, max score 100; the higher the score, the better the management of diabetes.
Nutrition diaries as assessed by a dietician | 0, 6 months
  Change in carbohydrates grams - baseline to 6 months. Assessment of carbohydrates in grams by a certified pediatric nutritionist.
Sleep quality as assessed by a questionnaire | 0, 6 months
  Change in sleep quality - baseline to 6 months, as assessed by a validated questionnaire, as cited in the Reference section.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Please Select, Israel

IPD SHARING:
Plan to Share IPD: Undecided
If requested, we will share the data collection system as needed.

REFERENCES:
- [Background] Mehta SN, Nansel TR, Volkening LK, Butler DA, Haynie DL, Laffel LM. Validation of a contemporary adherence measure for children with Type 1 diabetes: the Diabetes Management Questionnaire. Diabet Med. 2015 Sep;32(9):1232-8. doi: 10.1111/dme.12682. Epub 2015 Jan 30. PMID 26280463
- [Result] Skinner TC, Hoey H, McGee HM, Skovlund SE; Hvidore Study Group on Childhood Diabetes. A short form of the Diabetes Quality of Life for Youth questionnaire: exploratory and confirmatory analysis in a sample of 2,077 young people with type 1 diabetes mellitus. Diabetologia. 2006 Apr;49(4):621-8. doi: 10.1007/s00125-005-0124-0. Epub 2006 Jan 26. PMID 16525844
- [Result] Gaudry E, Vagg P, Spielberger CD. Validation of the State-Trait Distinction in Anxiety Research. Multivariate Behav Res. 1975 Jul 1;10(3):331-41. doi: 10.1207/s15327906mbr1003_6. PMID 26829634
- [Result] Gonder-Frederick L, Nyer M, Shepard JA, Vajda K, Clarke W. Assessing fear of hypoglycemia in children with Type 1 diabetes and their parents. Diabetes Manag (Lond). 2011;1(6):627-639. doi: 10.2217/DMT.11.60. PMID 22180760
- [Result] Rovner AJ, Nansel TR, Mehta SN, Higgins LA, Haynie DL, Laffel LM. Development and validation of the type 1 diabetes nutrition knowledge survey. Diabetes Care. 2012 Aug;35(8):1643-7. doi: 10.2337/dc11-2371. Epub 2012 Jun 4. PMID 22665217
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771